CLINICAL TRIAL: NCT04905199
Title: Bedside Precise Temporary Transvenous Cardiac Pacemaker Placement by Intracavitary Electrocardiogram Monitoring
Brief Title: Temporary Transvenous Pacemaker Placement by Intracavitary Electrocardiogram Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Meng Liu, Attending physician, Hunan Provincial People's Hospital
Other Study IDs: 202084
Record Dates: First submitted 2021-05-25; First posted 2021-05-27 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Bradycardia; Syncope; Bradyarrhythmia; Brady-tachy Syndrome; Tachycardia Bradycardia; AVB - Atrioventricular Block; Tachyarrhythmia
MeSH Terms: conditions — Bradycardia; Syncope; Atrioventricular Block; Tachycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-floating catheter: When using non-floating catheter.
  Interventions: Procedure: Temporary transvenous cardiac pacing
- Floating catheter: When using floating catheter.
  Interventions: Procedure: Temporary transvenous cardiac pacing

INTERVENTIONS:
Procedure: Temporary transvenous cardiac pacing — Transvenous temporary pacemaker insertion by modified IC-ECG monitoring.

SUMMARY:
Traditional temporary pacing catheter insertion by intracavitary electrocardiogram (IC-ECG) monitoring which only monitoring tip polar, the negative one. The investigators modified the technique by monitoring both negative and positive polar which will be precisely locating catheter tip and indicating the direction of the catheter tip.

Extensively used temporary pacing catheter tip has two electrodes which are about 1 cm apart. Distal electrode is negative (-) and active, proximal electrode is positive (+) and indifferent.

Investigators use both distal (-) and proximal (+) electrodes which can be attached to any two of the V leads, record as V(-) and V(+). Monitoring positions of the electrodes by V(-) and V(+) could provide more information about the tip position. Comparing the QRS amplitudes between V(-) and V(+), when catheter tip enters right ventricle chamber: the case of V(-) > V(+) infers tip toward apex ventricle wall ; conversely, the case of V(-)<V(+) indicates tip directs to outflow tract.

The investigators hypothesis this monitoring will help precisely placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of temporary transvenous pacing

Exclusion Criteria:

* Not applicate to IC-ECG monitoring.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients need emergency or selective temporary pacing.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Pacer leads location | One day.
  Satisfy location is in the apex of the right ventricle.
Catheter-related complications | One month.
  Pacing catheter related complications: tip dislocation caused pacemaker malfunction, myocardial injury, perforation, death.

SECONDARY OUTCOMES:
Other complications | One month.
  Complications not relate to pacing catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaotong Han, MD, Study Director — Hunan Provincial People's Hospital
Locations (1):
- Hunan Provincial People's hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Any date will share if appropriate.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Two years.